CLINICAL TRIAL: NCT04510805
Title: Single-blind, Randomized Comparison of Warfarin Management Guided by NextDose Versus Management Based on Clinician Experience.
Brief Title: Effectiveness of NextDose for Warfarin Dose Individualization
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Miao Liyan, vice-president, The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020025
Record Dates: First submitted 2020-08-11; First posted 2020-08-12 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Thrombosis Embolism
Keywords: warfarin; PKPD; Bayesian forecasting
MeSH Terms: conditions — Embolism and Thrombosis

STUDY DESIGN:
Intervention Model Description: Current warfarin dose individualization methods tend to be empirical, rather than based upon pharmacological and statistical principles. A theory-based model of warfarin pharmacokinetics and pharmacodynamics (PKPD) has been developed for dose individualization when used in conjunction with a Bayesian forecasting tool (NextDose).
  This study compares standard of care clinician judgement for warfarin management with the use of a web-based dosing tool (NextDose). Computer-assisted anticoagulant dosing has been shown to be helpful using empirical models. This study will evaluate a theory-based model which has shown superior performance over empirical models in predicting clinical doses of warfarin. The study is also guided by quality and service improvement principles.
Who Masked: Participant
Masking Description: All patients who are screened for enrolment will be allocated an enrolment number. The recruiting clinician will record into a logbook the details of all patients screened for enrolment, including the reason for exclusion from trial entry.
  A randomization sequence using block randomization with random block sizes of 4, 6 and 8 (to maintain equal sample size in each arm) will be created by researchers using PASS. Assignments will be enclosed in sequentially numbered, opaque, sealed envelopes.
  Participants who provide written informed consent and are enrolled will be allocated to study arm by the study pharmacists. The pharmacist will be responsible for opening envelopes sequentially, writing the participant enrollment number on the envelope prior to opening, and recording the envelope number and study arm allocation in the CRF. On conclusion of the data collection phase, the (actual) study allocation status of the participants will be compared to the randomization sequence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): NextDose guided warfarin management taking into consideration covariates (sex, age, weight, height CYP2C9 (rs1057910) and VKORC1 (rs9923231), the dosing and INR history of each patient to predict an individualized dose in accordance with the theory-based warfarin model and target concentration intervention principles.
  Initial recommended warfarin dose, up to the first INR, will be the maintenance dose predicted from group values, subsequently the NextDose predicted maintenance dose will be recommended. The treating clinician will also be provided with the NextDose report to inform the choice of the prescribed dose.
  Interventions: Device: NextDose (nextdose.org)
- Control Arm (No Intervention): Usual standard of care. Clinical experience of the treating physician taking into account the covariates, dosing and INR history of each patient, to determine the initial, and subsequent maintenance doses.

INTERVENTIONS:
Device: NextDose (nextdose.org) — NextDose guided warfarin management taking into consideration covariates (sex, age, weight, height CYP2C9 (rs1057910) and VKORC1 (rs9923231), the dosing and INR history of each patient to predict an individualized dose in accordance with the theory-based warfarin model and target concentration intervention principles.
  Initial recommended warfarin dose, up to the first INR, will be the maintenance dose predicted from group values, subsequently the NextDose predicted maintenance dose will be recommended. The treating clinician will also be provided with the NextDose report to inform the choice of the prescribed dose.
  Arms: Intervention Arm

SUMMARY:
Objectives:

To understand whether the implementation of warfarin dose management using NextDose (nextdose.org) at The First Affiliated Hospital of Soochow University (Suzhou, China) improves the quality of anticoagulation therapy.

Endpoint Primary

1. Percentage of time within the acceptable INR range estimated using linear interpolation during the 28 days after initiation of warfarin.

Secondary 2.1 Percentage of Time Measures 2.2 Time to Stable Dose 2.3 Safety Outcomes 2.4 Acceptability of NextDose Recommendations Exploratory 3.1 Percentage of Time Measures 3.2 Time to Stable Dose 3.3 Safety Outcomes 3.4 Acceptability of NextDose Recommendations 3.5 Model Evaluation 3.6 INR Variability

Population:

240 participants of any sex between the age of 18 and 80 years. Patients requiring treatment with warfarin following cardiac surgery.

DETAILED DESCRIPTION:
Objectives:

To understand whether the implementation of warfarin dose management using NextDose (nextdose.org) at The First Affiliated Hospital of Soochow University (Suzhou, China) improves the quality of anticoagulation therapy.

Endpoint Primary

1. Percentage of time within the acceptable INR range estimated using linear interpolation during the 28 days after initiation of warfarin.

   Secondary 2.1 Percentage of Time Measures
   1. Percentage of time within the acceptable INR Range estimated using linear interpolation during the 90 days after initiation of warfarin.
   2. Percentage of time spent above and below the acceptable INR range at day 28, and 90 after initiation of warfarin estimated by linear interpolation.

   2.2 Time to Stable Dose a. Number of days to achievement of stable dose (defined as 3 consecutive INR measurements within acceptable range for the same mean daily dose).

   2.3 Safety Outcomes a. Number of participants who experience at least one of the following safety events: major bleeding within 30 days, INR of 4 or greater within 30 days, death within 30 days, and symptomatic or asymptomatic VTE confirmed by objective testing within 60 days of surgery.

   2.4 Acceptability of NextDose Recommendations
   1. Percentage of prescribed doses within 0.625 mg of the NextDose proposed dose.
   2. Mean difference between the prescribed dose and the NextDose proposed dose. Exploratory 3.1 Percentage of Time Measures

   a. The percentage of time spent within, above and below the acceptable INR range estimated by numerical integration with the Bayesian parameter estimates of the PKPD model at day 28 and at day 90 after initiation of warfarin.

   3.2 Time to Stable Dose a) Days to first INR measurement within the acceptable range. b) Days to second consecutive INR measurement within the acceptable range. c) Number of dose adjustments to achievement of stable dose (3 consecutive INR measurements within acceptable range for the same mean daily dose).

   d) Total number of dose adjustments at day 90. e) Total number of INR measurements at day 90. 3.3 Safety Outcomes

   a) Incidence of minor and major bleeding events. b) Incidence of thromboembolic events. c) 30 day all-cause mortality. d) 90 day all-cause mortality. e) 90 day cardiovascular mortality. f) Number of warfarin doses withheld due to high INR (as determined by the treating clinician).

   3.4 Acceptability of NextDose Recommendations a) Percentage of prescribed doses within 20% of the NextDose proposed dose. 3.5 Model Evaluation

   a) Predictive performance of the model for patients with steady-state warfarin doses below 2 or above 7 mg/day.

   3.6 INR Variability

   a) INR variability as described by Lind et al. (the standard deviation of transformed INR values).

   Population:

240 participants of any sex between the age of 18 and 80 years. Patients requiring treatment with warfarin following cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo cardiac surgery with planned warfarin anticoagulation for at least three months.
* Age ≥ 18 and < 80 years.
* Written informed consent has been obtained.

Exclusion Criteria:

* Allergy to warfarin tablet or excipients.
* Enrollment or planned enrollment in other research that would conflict with full participation in the study or confound the observation or interpretation of the study findings.
* Patients who in the opinion of the recruiting clinician are:

  * unwilling or unable to comply with the protocol requirements and/or,
  * considered unreliable concerning the requirements for follow-up during the study and/or, compliance with drug administration.
* Patient with life expectancy less than the expected duration of the trial due to concomitant disease.
* Contraindication to warfarin therapy. The following are examples but not an exhaustive list:

  * Pregnancy.
  * Cerebral infarction or cerebral haemorrhage (from patients' medical record) within the 3 months prior to heart valve replacement
  * Severe heart failure (New York Heart Function Class IV)
  * Severe renal failure (CLcr (Cockcroft-Gault) ≤20mL / min)
  * Severe liver failure (Child-Pugh≥10)
  * Abnormal liver function (elevated transaminase more than three times the upper limit of the local hospital clinical laboratory).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Time Within Range | 28 days after initiation of warfarin
  The percentage of time spent within the acceptable INR range (± 0.5 of target INR) as estimated using linear interpolation during the 28 days after initiation of warfarin.

SECONDARY OUTCOMES:
Percentage of Time Measure | day 90 after initiation of warfarin
  The percentage of time spent within the acceptable INR range at day 90 after initiation of warfarin estimated by linear interpolation.
Percentage of Time Measure | day 28, and 90 after initiation of warfarin
  The percentage of time spent above and below the acceptable INR range at day 28, and 90 after initiation of warfarin estimated by linear interpolation.
Time to Stable Dose | 90 days after initiation of warfarin
  Number of days to achievement of stable dose (defined as 3 consecutive INR measurements within acceptable range for the same mean daily dose.
Number of participants who experience at least one of the following safety events: | 60 days of surgery.
  major bleeding within 30 days, INR of 4 or greater within 30 days, death within 30 days, and symptomatic or asymptomatic VTE confirmed by objective testing within 60 days of surgery.
Percentage of prescribed doses within 0.625 mg of the NextDose proposed dose. | 90 days after initiation of warfarin
  Acceptability of NextDose Recommendations
Mean difference between the prescribed dose and the NextDose proposed dose. | 90 days after initiation of warfarin
  Acceptability of NextDose Recommendations

CONTACTS AND LOCATIONS:
Overall Officials: Li Y Miao, PhD, Principal Investigator — The First Affiliated Hospital of Soochow University; Zhen Y Shen, PhD, Principal Investigator — The First Affiliated Hospital of Soochow University; Nick Holford, MBChB, Study Director — University of Auckland, New Zealand; Ling Xue, MS, Study Director — The First Affiliated Hospital of Soochow University; Guangda Ma, MHSc, Study Director — University of Auckland, New Zealand; Ying L Ding, MS, Study Director — The First Affiliated Hospital of Soochow University; Qiong Qin, MS, Study Director — The First Affiliated Hospital of Soochow University; Jacqui Hannam, PhD, Study Director — University of Auckland, New Zealand

REFERENCES:
- [Result] Sheiner LB. Computer-aided long-term anticoagulation therapy. Comput Biomed Res. 1969 Dec;2(6):507-18. doi: 10.1016/0010-4809(69)90030-5. No abstract available. PMID 5367362
- [Result] Boyle DA, Ludden TM, Carter BL, Becker AJ, Taylor JW. Evaluation of a Bayesian regression program for predicting warfarin response. Ther Drug Monit. 1989;11(3):276-84. doi: 10.1097/00007691-198905000-00010. PMID 2728086
- [Result] Xue L, Holford N, Ding XL, Shen ZY, Huang CR, Zhang H, Zhang JJ, Guo ZN, Xie C, Zhou L, Chen ZY, Liu LS, Miao LY. Theory-based pharmacokinetics and pharmacodynamics of S- and R-warfarin and effects on international normalized ratio: influence of body size, composition and genotype in cardiac surgery patients. Br J Clin Pharmacol. 2017 Apr;83(4):823-835. doi: 10.1111/bcp.13157. Epub 2016 Nov 25. PMID 27763679
- [Result] Higashi MK, Veenstra DL, Kondo LM, Wittkowsky AK, Srinouanprachanh SL, Farin FM, Rettie AE. Association between CYP2C9 genetic variants and anticoagulation-related outcomes during warfarin therapy. JAMA. 2002 Apr 3;287(13):1690-8. doi: 10.1001/jama.287.13.1690. PMID 11926893
- [Result] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Result] Leon MB, Piazza N, Nikolsky E, Blackstone EH, Cutlip DE, Kappetein AP, Krucoff MW, Mack M, Mehran R, Miller C, Morel MA, Petersen J, Popma JJ, Takkenberg JJ, Vahanian A, van Es GA, Vranckx P, Webb JG, Windecker S, Serruys PW. Standardized endpoint definitions for Transcatheter Aortic Valve Implantation clinical trials: a consensus report from the Valve Academic Research Consortium. J Am Coll Cardiol. 2011 Jan 18;57(3):253-69. doi: 10.1016/j.jacc.2010.12.005. Epub 2011 Jan 7. PMID 21216553
- [Derived] Xue L, Ma G, Holford N, Qin Q, Ding Y, Hannam JA, Ding X, Fan H, Ji Z, Yang B, Shen H, Shen Z, Miao L. A Randomized Trial Comparing Standard of Care to Bayesian Warfarin Dose Individualization. Clin Pharmacol Ther. 2024 Jun;115(6):1316-1325. doi: 10.1002/cpt.3207. Epub 2024 Mar 4. PMID 38439157
- See also: NextDose — https://www.nextdose.org/